CLINICAL TRIAL: NCT00933530
Title: A Phase I Randomized, Placebo-Controlled, Single-Blind, Multiple-Dose, Dose-Escalation Clinical Study to Assess the Safety and Pharmacokinetics of SRT2104 in Normal Healthy Male Volunteers
Brief Title: A Clinical Study to Assess the Safety and Pharmacokinetics of SRT2104 in Normal Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 113259
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2; Healthy Volunteer
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 - Dose Level A (0.03g/day) (Experimental): 0.03g SRT2104 dosing will take place at approximately the same time every morning after fasting for at least 10 hours. Subjects will be required to stay overnight at the study center for all dosing days. Six subjects are assigned to this cohort. On Day1 of the single dosing period, one subject will be dosed with 0.03g SRT2014 while one is dosed with placebo on Day1. If no safety issues arise from this dosing, then on Day2, three subjects will be dosed with 0.03g SRT2104 while one is dosed with placebo. Subjects within the cohort will remain on a fixed dose for all dosing days.
  This cohort of subjects will be dosed sequentially approximately two weeks apart from the single dose period, and return to the clinic approximately one week after their single dose administration to receive 7 consecutive days of daily dosing for the multiple dose period. A comprehensive safety assessment will be conducted one week prior to the initiation of an escalated dose in the subsequent cohort.
  Interventions: Drug: SRT2104; Drug: Placebo
- Cohort 2 - Dose Level B (0.1g/day) (Experimental): 0.1g SRT2104 dosing will take place at approximately the same time every morning after fasting for at least 10 hours. Subjects will be required to stay overnight at the study center for all dosing days. Six subjects are assigned to this cohort. On Day1 of the single dosing period, one subject will be dosed with 0.1g SRT2014 while one is dosed with placebo on Day1. If no safety issues arise from this dosing, then on Day2, three subjects will be dosed with 0.1g SRT2104 while one is dosed with placebo. Subjects within the cohort will remain on a fixed dose for all dosing days.
  This cohort of subjects will be dosed sequentially approximately two weeks apart from the single dose period, and return to the clinic approximately one week after their single dose administration to receive 7 consecutive days of daily dosing for the multiple dose period. A comprehensive safety assessment will be conducted one week prior to the initiation of an escalated dose in the subsequent cohort.
  Interventions: Drug: SRT2104; Drug: Placebo
- Cohort 3 - Dose Level C (0.25g/day) (Experimental): 0.25g SRT2104 dosing will take place at approximately the same time every morning after fasting for at least 10 hours. Subjects will be required to stay overnight at the study center for all dosing days. Six subjects are assigned to this cohort. On Day1 of the single dosing period, one subject will be dosed with 0.25g SRT2014 while one is dosed with placebo on Day1. If no safety issues arise from this dosing, then on Day2, three subjects will be dosed with 0.25g SRT2104 while one is dosed with placebo. Subjects within the cohort will remain on a fixed dose for all dosing days.
  This cohort of subjects will be dosed sequentially approximately two weeks apart from the single dose period, and return to the clinic approximately one week after their single dose administration to receive 7 consecutive days of daily dosing for the multiple dose period. A comprehensive safety assessment will be conducted one week prior to the initiation of an escalated dose in the subsequent cohort.
  Interventions: Drug: SRT2104; Drug: Placebo
- Cohort 4 - Dose Level D (0.5g/day) (Experimental): 0.5g SRT2104 dosing will take place at approximately the same time every morning after fasting for at least 10 hours. Subjects will be required to stay overnight at the study center for all dosing days. Six subjects are assigned to this cohort. On Day1 of the single dosing period, one subject will be dosed with 0.5g SRT2014 while one is dosed with placebo on Day1. If no safety issues arise from this dosing, then on Day2, three subjects will be dosed with 0.5g SRT2104 while one is dosed with placebo. Subjects within the cohort will remain on a fixed dose for all dosing days.
  This cohort of subjects will be dosed sequentially approximately two weeks apart from the single dose period, and return to the clinic approximately one week after their single dose administration to receive 7 consecutive days of daily dosing for the multiple dose period. A comprehensive safety assessment will be conducted one week prior to the initiation of an escalated dose in the subsequent cohort.
  Interventions: Drug: SRT2104; Drug: Placebo
- Cohort 5 - Dose Level E (1.0g/day) (Experimental): 1.0g SRT2104 dosing will take place at approximately the same time every morning after fasting for at least 10 hours. Subjects will be required to stay overnight at the study center for all dosing days. Six subjects are assigned to this cohort. On Day1 of the single dosing period, one subject will be dosed with 1.0g SRT2014 while one is dosed with placebo on Day1. If no safety issues arise from this dosing, then on Day2, three subjects will be dosed with 1.0g SRT2104 while one is dosed with placebo. Subjects within the cohort will remain on a fixed dose for all dosing days.
  This cohort of subjects will be dosed sequentially approximately two weeks apart from the single dose period, and return to the clinic approximately one week after their single dose administration to receive 7 consecutive days of daily dosing for the multiple dose period. A comprehensive safety assessment will be conducted one week prior to the initiation of an escalated dose in the subsequent cohort.
  Interventions: Drug: SRT2104; Drug: Placebo
- Cohort 6 - Dose Level F (2.0g/day) (Experimental): 2.0g SRT2104 dosing will take place at approximately the same time every morning after fasting for at least 10 hours. Subjects will be required to stay overnight at the study center for all dosing days. Six subjects are assigned to this cohort. On Day1 of the single dosing period, one subject will be dosed with 2.0g SRT2014 while one is dosed with placebo on Day1. If no safety issues arise from this dosing, then on Day2, three subjects will be dosed with 2.0g SRT2104 while one is dosed with placebo. Subjects within the cohort will remain on a fixed dose for all dosing days.
  This cohort of subjects will be dosed sequentially approximately two weeks apart from the single dose period, and return to the clinic approximately one week after their single dose administration to receive 7 consecutive days of daily dosing for the multiple dose period. A comprehensive safety assessment will be conducted one week prior to the initiation of an escalated dose in the subsequent cohort.
  Interventions: Drug: SRT2104; Drug: Placebo
- Cohort 7 - Dose Level G (3.0g/day) (Experimental): 3.0g SRT2104 dosing will take place at approximately the same time every morning after fasting for at least 10 hours. Subjects will be required to stay overnight at the study center for all dosing days. Six subjects are assigned to this cohort. On Day1 of the single dosing period, one subject will be dosed with 3.0g SRT2014 while one is dosed with placebo on Day1. If no safety issues arise from this dosing, then on Day2, three subjects will be dosed with 3.0g SRT2104 while one is dosed with placebo. Subjects within the cohort will remain on a fixed dose for all dosing days.
  This cohort of subjects will be dosed sequentially approximately two weeks apart from the single dose period, and return to the clinic approximately one week after their single dose administration to receive 7 consecutive days of daily dosing for the multiple dose period.
  Interventions: Drug: SRT2104; Drug: Placebo

INTERVENTIONS:
Drug: SRT2104 — SRT2104 (0.03, 0.1, 0.25, 0.5, 1.0, 2.0, or 3.0 g/day) will be supplied as a powder which will be prepared by the Pharmacist/designee into a liquid suspension. The dosing vehicle is 1% (by weight) hypromellose acetate succinate in water, which is used as a suspension aid and a dispersant for the SRT2104. Test material will be administered orally, in a single dose and subsequently, once daily for seven consecutive days. A trained staff member will prepare individual solutions of test material that the subject will drink once daily in the clinic following a 10-hour (minimum) fast.
  Other Names: GSK2245840
Drug: Placebo — Placebo (at the matched dosage as SRT2104) will be supplied as a powder which will be prepared by the Pharmacist/designee into a liquid suspension. Placebo will consist of titanium dioxide USP and prepared for oral administration identically to the SRT2104 investigational product. Test material will be administered orally, in a single dose and subsequently, once daily for seven consecutive days. The subjects enrolled will be blinded to treatment assignment. A trained staff member will prepare individual solutions of test material that the subject will drink once daily in the clinic following a 10-hour (minimum) fast.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of SRT2104 (0.03, 0.1, 0.25, 0.5, 1.0, 2.0, and 3.0 g/day) in healthy male volunteers when administered after a single dose and once daily for 7 consecutive days.

The purpose is also to characterize the pharmacokinetic profile of SRT2104 (0.03, 0.1, 0.25, 0.5, 1.0, 2.0, and 3.0 g/day) after a single dose and multiple administrations in healthy male volunteers.

DETAILED DESCRIPTION:
Prospective, single center, clinical study of SRT2104 administered orally. Randomized, placebo-controlled, single-blind, multiple-dose, dose-escalation inpatient/outpatient study to assess the safety and pharmacokinetics (PK) of SRT2104 in healthy male volunteers. Forty-two (42) subjects aged 18-55, who fulfill the inclusion/exclusion criteria, will be enrolled in this study. Seven cohorts of six subjects each will be examined. Subjects within each cohort will be randomized 4:2 to receive SRT2104 at one of seven escalating doses (A, B, C, D, E, F, or G), likely to be 0.03, 0.1, 0.25, 0.5, 1.0, 2.0, or 3.0 g/day or placebo. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving active treatment and one subject receiving placebo. The remainder of subjects within each cohort will be dosed on Day 2 of the single dose period with three subjects receiving active treatment and one subject receiving placebo assuming that no safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study.

Each cohort of subjects will be dosed sequentially approximately two weeks apart for the single dose period, and return to the clinic approximately one week after their single dose administration to receive 7 consecutive days of dosing for the multiple dose period. Each cohort of subjects in the multiple dose period will be dosed sequentially, approximately, one week apart, allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort. In the event of suspected drug related toxicity, as determined by the principal investigator, sponsor, and an independent medical monitor, at a dose of 0.03 g/day, all subjects in the 0.03 g/day cohort will discontinue dosing, and the subsequent cohort will receive 0.01 g/day for seven consecutive days. Safety and PK-related data will be reviewed for the 0.01 g/day dose level, and no subsequent cohorts will be enrolled into the study.

Subjects will sign the informed consent form at the screening visit. If eligible and willing to participate, subjects will enter into the study. Subjects will have fasted for at least 10 hours overnight and be randomized to receive SRT2104 or placebo (test material). Subjects will be required to stay overnight at the study center for two nights during the single dose period of the study and subsequently, for the duration of the seven-day multiple dose period to assess safety and to gather required PK samples. Subjects will be asked to return to the study center for an End of Study safety assessment 1 week after they complete the multiple dose period.

Dose escalation will be dependent on safety parameters (physical examination findings, vital signs, ECG studies, adverse events and laboratory values) and PK data.

ELIGIBILITY:
Inclusion Criteria:

* Be male within the age range of 18 to 55 years.
* Voluntarily sign an Independent Review Board (IRB/IEC)-approved informed consent form to participate in the study after all relevant aspects of the study have been explained and discussed with the subject.
* Have Hematology, Coagulation, Clinical Chemistry and Urinalysis test results that are within normal, allowable limits (if out-of-range, must be considered clinically significant to be exclusionary) and performed within 21 days of receiving first dose of test material.
* Have a BMI (Body Mass Index) between 18.0 and 30.0 kg/m2.
* Be clear of any history of HIV 1 and 2 and hepatitis B and C.
* Have no significant disease or clinically significant abnormal laboratory value as deemed by the investigator on the laboratory evaluations, medical history, or physical exam.
* Have a normal 12-lead ECG or an ECG with abnormality considered to be clinically insignificant.
* Have the ability to communicate with the investigative site staff in a manner sufficient to carry out all protocol procedures as described.
* Subject and their partner must agree to use an acceptable double barrier method for birth control from the Screening visit through 3 months after the last dose of test material.
* Subject agrees to refrain from consumption of grapefruits and/or grapefruit juice from time of study enrollment through end of subject's final study visit.

Exclusion Criteria:

* Subject has had a major illness in the past three months or any significant ongoing chronic medical illness that the Investigator would deem unfavorable for enrollment.
* Subject has renal or liver impairment.
* Subject has a history of gastro-intestinal surgery or has a current gastrointestinal disease which may influence drug absorption.
* Subject has a history, within 3 years, of drug abuse (including Benzodiazepines, opioids, amphetamine, cocaine, and THC) or a positive drug result at Screening.
* Subject has a history of smoking, within 3 months, or is currently a smoker.
* Subject has a history of alcoholism (more than two years), and/or is currently drinking more than three drinks per day [one drink is equal to one unit of alcohol (one glass of wine, half a pint of beer, one measure of a spirit)].
* Subject has participated in a clinical trial within the past three months.
* Subject has a history of difficulty in donating blood or accessibility of veins in left or right arm.
* Subject has donated blood (one unit or 350 mL) within three months prior to receiving test material.
* Subject is taking herbal products or prescription drug therapy for which 5 times the half-life is longer than 21 days (i.e., the Screening period) prior to enrollment into the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SRT2104 (0.03, 0.1, 0.25, 0.5, 1.0, 2.0, and 3.0 g/day) when administered as a single dose and when administered once daily for 7 consecutive days. | Adverse events will be monitored continuously while subjects are on study; safety visits will occur every 7 days for the duration of subject participation.
Characterize the pharmacokinetic profile of SRT2104 (0.03, 0.1, 0.25, 0.5, 1.0, 2.0, and 3.0 g/day) when administered as a single dose and when administered as once daily for 7 consecutive days. | Single dose PK timepoints are: predose and 15min, 30min, 1h, 2h, 4h, 8h, 12h, 24hrs postdose. Multiple dose PK timepoints are: Day1 to Day6 predose, Day7 predose, and 15min, 30min, 1h, 2h, 4h, 8h, 12h, 24hrs postdose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Merthyr Tydfill, Glamorgan, United Kingdom